CLINICAL TRIAL: NCT00187720
Title: Genetic Basis for Variation in the Renal Elimination of Metformin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 787
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2012-12

CONDITIONS: Other Conditions That May Be A Focus of Clinical Attention
Keywords: Healthy Control
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OCT2-variant Group (Experimental): Subjects with OCT2-variant genotype will be given a single oral dose of 850 mg of metformin.
  Interventions: Drug: Metformin
- OCT2-reference Group (Experimental): Subjects with OCT2-reference genotype will be given a single oral dose of 850 mg of metformin.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Subjects will be given a single oral dose of 850 mg of metformin
  Other Names: GLUCOPHAGE

SUMMARY:
The current study is part of a large multi-investigator grant to look at the pharmacogenetics of a number of membrane transporters. We will study individuals with particular genotypes of the human organic cation transporter, (hOCT2), to test the hypothesis that genetic variation in hOCT2 is associated with variation in the renal clearance of the antidiabetic agent, metformin.

DETAILED DESCRIPTION:
The drug, which is used in the treatment of Type II diabetes, has a narrow therapeutic range. Its net renal clearance by secretion (i.e., renal clearance minus filtration clearance) ranges from approximately 100 ml/min to 800ml/min in normal, healthy subjects. Although many factors may contribute to inter-individual variation in renal secretory clearance, initial estimates of heritability (greater than 0.6) suggest that genetic factors play an important role in the renal secretion of metformin. Available evidence supports the idea that hOCT2 is the primary transporter involved in the first-step of renal secretion of metformin, i.e., uptake from the blood to the tubule cell across the basolateral membrane. In particular, (a) hOCT2 is the primary organic cation transporter on the basolateral membrane of the human kidney; and (b) metformin interacts with and is translocated by hOCT2 in heterologous expression systems.

In recent studies, we identified four variants (M165I, A270S, R400C, and K432Q) with ethnic-specific allele frequencies ≥1% [6] that have altered function in studies in heterologous expression systems. In addition, we identified a common haplotype of hOCT2 and one haplotype that contain the non-synonymous cSNP, A270S. We will determine whether variability in the renal secretory clearance of the model organic cation, metformin, in healthy individuals is associated with genetic variation in hOCT2. In particular, we will determine whether the renal clearance of metformin differs in individuals who are homozygous for the common haplotype of OCT2 (OCT2*1) and those who are heterozygous for the less common haplotype OCT2*3D, which we have identified in a comprehensive screen of ethnically identified DNA samples. We will also determine whether individuals who are heterozygous for the less common OCT2 variants, M165I, R400C and K432Q, have reduced renal clearances of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have previously participated in the Study Of Pharmacogenetics In Ethnically Diverse Populations (SOPHIE) study.
* 18-40 years old
* Possess a pre-specified genotype for OCT2

Exclusion Criteria:

* Taking any regular medications other than vitamins.
* Individuals with anemia (hemoglobin < 12 g/dL), an elevation in liver enzymes to higher than double the respective normal value, or elevated creatinine concentrations (males ≥ 1.5 mg/dL, females ≥ 1.4 mg/dL)
* Pregnant or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2002-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Giacomini, PhD, Principal Investigator — University of California, San Francsico
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Result] Chen Y, Li S, Brown C, Cheatham S, Castro RA, Leabman MK, Urban TJ, Chen L, Yee SW, Choi JH, Huang Y, Brett CM, Burchard EG, Giacomini KM. Effect of genetic variation in the organic cation transporter 2 on the renal elimination of metformin. Pharmacogenet Genomics. 2009 Jul;19(7):497-504. doi: 10.1097/FPC.0b013e32832cc7e9. PMID 19483665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment were 5/2003 through 4/10/2007. Location was General Clinical Research Center (GCRC) at San Francisco General Hospital.
Groups:
- Organic Cation Transporter 2 (OCT2)-Variant Group: Subjects with OCT2-variant genotype will be given a single oral dose of 850 mg of metformin
- Organic Cation Transporter 2 (OCT2)-Reference Group: Subjects with OCT2-reference genotype will be given a single oral dose of 850 mg of metformin
Period: Overall Study
Arm/Group | Organic Cation Transporter 2 (OCT2)-Variant Group | Organic Cation Transporter 2 (OCT2)-Reference Group
Started | 9 | 14
Completed | 9 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OCT2-reference Group | OCT2-variant Group | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 9 | 23
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.3 (6.6) | 31.2 (5.5) | 28.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 14 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Renal Clearance of Metformin
Description: To test whether individuals with genetic variants of the human organic cation transporter, OCT2, exhibit altered renal elimination of metformin we will measure the difference in renal clearance between reference and variant groups.
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours
Population: Analysis was per protocol. The sample size of 23 subjects will enable us to detect a significant difference (at the p < 0.05 level; α = 0.05, β = 0.80) in the renal clearance of metformin between individuals who are homozygous for the reference OCT2 and those who carry the OCT2 variant A270S allele.
Measure: Mean (Standard Deviation); unit: mL/min
Groups:
- OCT2-variant Group: The renal clearance of metformin in subjects heterozygous for the variant OCT2 genotype (808G/T, *3D) following a single oral dose of 850 mg of metformin.
- OCT2-reference Group: The renal clearance of metformin in subjects homozygous for the reference OCT2 genotype (808G/G) following a single oral dose of 850 mg of metformin.
Arm/Group | OCT2-variant Group | OCT2-reference Group
Number analyzed (Participants) | 9 | 14
mL/min | 614 (158) | 441 (108)

ADVERSE EVENTS:
Arm/Group | OCT2-reference Group | OCT2-variant Group
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/9
Other Adverse Events (participants affected / at risk) | 0/14 | 0/9

LIMITATIONS AND CAVEATS:
Recruitment of subjects with interested genotypes was our limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No